CLINICAL TRIAL: NCT00178282
Title: Pilot Study: Low Intensity Physical Therapy for Prevention of Pre and Postpartum Urinary Incontinence
Brief Title: Low-Intensity Physical Therapy for Prevention of Pre and Postpartum Urinary Incontinence
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated early due to poor subject enrollment.
Sponsor: University of Rochester (Other)
Collaborators: Watson Pharmaceuticals (Industry)
Responsible Party: Gunhilde Buchsbaum, MD, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11098
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2011-11-03 (Estimated); Status verified 2011-11

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Pelvic Floor Muscle exercises

SUMMARY:
The purpose of this study is to determine if pelvic exercises can reduce the occurrence of urinary incontinence (involuntary loss of urine) before and after delivery. We would also like to see if performing pelvic exercises before birth has an effect on labor and/or delivery, and if there are any specific characteristics for developing urinary incontinence during pregnancy and after delivery.

DETAILED DESCRIPTION:
The studies investigating physiotherapy for prevention of urinary incontinence during and after pregnancy used intensive pelvic floor muscle training. While physical therapy appears to be effective in preventing urinary incontinence, extensive physical therapy is too costly to be implemented as a preventive measure for the general population. Thus, we want to asses if non-intensive pelvic floor therapy decreases the urinary incidence of incontinence during pregnancy and postpartum. We propose a prospective randomized controlled trial to obtain baseline data on the effect of non-intensive pelvic floor muscle training of urinary incontinence in primigravid women.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous, pregnant women, 18 years or older
* Less than 20 weeks gestation
* Able to give consent and who are willing to participate

Exclusion Criteria:

* Multiparous women
* Women presenting after 20 weeks gestation
* History of urinary incontinence
* Mentally impaired women and women who have neurological impairment affecting ability to perform pelvic floor muscle training

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-06; Primary Completion 2007-01 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Non-intensive physical therapy, 24hr. voiding diary, pad weight, Quality of Life questionnaires | During and 3 months after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Gunhilde Buchsbaum, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States